CLINICAL TRIAL: NCT04520646
Title: A Pilot Study of Empagliflozin in the Treatment of Acromegalic Cardiomyopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhaoyun Zhang, vice director of endocrine department, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2020-849
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Acromegaly; Cardiomyopathies
MeSH Terms: conditions — Acromegaly; Cardiomyopathies | interventions — empagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- empagliflozin (Experimental): empagliflozin is added on the basis of the original treatment
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — empagliflozin of 10mg/day is added on the basis of primary care

SUMMARY:
Acromegaly is a disease characterized by excess growth hormone(GH) and insulin like growth factor(IGF)-1. Pituitary GH secreting adenoma is the major cause of acromegaly. Acromegalic cardiomyopathy is one of the leading causes of death in acromegalic patients. No efficient medicine is available for acromegalic cardiomyopathy until now and there were limited studies. Empagliflozin is proved to decrease the risk of heart failure in diabetic patients and independent of blood glucose control. We planed to evaluate the structure of heart by MRI before and after 6 months treatment with empagliflozin in acromegalic patients to investigate the effect of empagliflozin on acromegalic cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* patients with pituitary GH adenomas confirmed by surgery

active acromegalic patients although treated with surgery,radiation therapy and somatostatin analogs

Exclusion Criteria:

* patients with contraindications to empagliflozin pregnant patients patients with poor control of hypertension(SBP>150mmHg or DBP>95mmHg patients with contraindications to MRI

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular mass index | 6 months
  the changes in left ventricular mass index by heart MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China